CLINICAL TRIAL: NCT04867512
Title: The Effects of a Botanical Blend on the Gut Microbiome and Gut-Skin-Axis in Small Intestinal Bacterial Overgrowth (SIBO)
Brief Title: Botanical Blend on the Gut Microbiome and Gut-Skin-Axis in Small Intestinal Bacterial Overgrowth (SIBO)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Integrative Skin Science and Research (Industry)
Collaborators: Biocidin (Unknown)
Responsible Party: Principal Investigator, Raja Sivamani, Principal Investigator, Integrative Skin Science and Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIOSIBO1
Record Dates: First submitted 2021-04-27; First posted 2021-04-30 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Small Intestinal Bacterial Overgrowth (SIBO)
Keywords: Small Intestinal Bacterial Overgrowth (SIBO); gut health; microbiome; skin; dermatology; botanical medicine

STUDY DESIGN:
Intervention Model Description: Open-Label Prospective Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): Participants will be taking one liquid tincture orally per day as well as 2 capsules orally at night. At week 10, non-responders will take another supplement consisting of 2 capsules orally along with the liquid tincture until week 14.
  Interventions: Dietary Supplement: Liquid Tincture; Dietary Supplement: GI Detox; Dietary Supplement: Olivirex

INTERVENTIONS:
Dietary Supplement: Liquid Tincture — Biocidin Liquid Tincture: 1 drop by mouth twice daily, increased by one drop each day until 15 drops twice daily have been reached. 15 drops by mouth twice daily will be maintained through the duration of the study.
Dietary Supplement: GI Detox — GI Detox: 2 capsules by mouth every evening and 1 hour away from all food maintained through the duration of the study.
Dietary Supplement: Olivirex — Olivirex: 2 capsules by mouth twice daily taken with Biocidin liquid tincture starting at week 10 until week 14 of the study for non-responders determined by symptoms and lactulose breath test results.

SUMMARY:
The purpose of this study is to assess how an oral botanical blend alters the gut microbiome and the skin biophysical properties in people with SIBO.

DETAILED DESCRIPTION:
Certain oral botanical blends have many antimicrobial properties. This study will evaluate if a botanical blend can improve the gut and skin health of people with small intestinal bacterial overgrowth (SIBO) since it is caused by an overgrowth of bacteria in the small intestine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 18-60 years of age
* Must be willing to comply with all protocol requirements
* Must be willing to have flash photo facial images taken with the imaging systems
* Males must be willing to shave any facial hair
* Subjects with (Small Intestine Bacterial Overgrowth) SIBO

Exclusion Criteria:

* Any systemic or antibiotics (injected or oral) within 6 months of starting the study.
* Any topical antibiotic or benzoyl peroxide within 2 months of starting the study or any subject unwilling to refrain from washout of topical antibacterial or benzoyl peroxide ingredient.
* Any other topical products within 2 weeks of starting the study.
* Any oral probiotics or prebiotics within 3 months of starting the study.
* Any other oral supplements within 3 months of starting the study.
* Subjects must have no history of malignancy or cancer or diagnosis of gastrointestinal inflammatory diseases, no history or diagnosis of epilepsy, no history or diagnosis of immunologic or infectious disease (e.g. hepatitis, tuberculosis, HIV or AIDS, lupus, rheumatoid arthritis, irritable bowel disease, multiple sclerosis, Parkinson's disease)
* Has a condition or is on medication the investigator and/or designee believe could jeopardize the safety of the subject, interfere with the evaluation, or confound the interpretation of the study results
* Has a condition where evening medication dosing is required
* Has any gastrointestinal motility condition
* Women who have been pregnant in the last three months, are pregnant, preparing to be pregnant or lactating, or post-menopausal.
* Is participating in a concurrent clinical research study or has participated in an acne or other facial study at this or any other facility in the past 4 weeks.
* Those with BMI higher than 35 kg/m².
* Commencement of a new diet (such as the ketogenic diet) or supplements within the 1 month prior to initiating participation, at the discretion of the investigator.
* Use of medications that alter blood lipids, such as statins and anti- hyperlipidemic medications.
* Is participating in or has participated in a facial study at this or any other facility in the past 4 weeks. Participation in survey-based studies is approved at the discretion of the investigator.
* Has a skin disease on face that will interfere with image collection and assessment in the opinion of the investigator.
* Refusal to shave or remove facial hair that may interfere with image collection and assessment.
* Persons unwilling to avoid the following during the 4 weeks prior and during the duration of the study: self-tanning, spa tanning, sun tanning, or artificial tanning.
* Known allergy or irritation to the facial products utilized in the study.
* Current tobacco smokers, OR those that have smoked tobacco over the past year, OR a 5 year-pack year history of smoking tobacco.
* Prisoners
* Any persons with current or a history of alcohol abuse
* Adults unable to consent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-04-27 (Estimated); Primary Completion 2021-04-30 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Lactulose Breath Test | 10 weeks
  Presence of SIBO
Lactulose Breath Test | 14 weeks
  Presence of SIBO

SECONDARY OUTCOMES:
Gut Microbiome Changes | 10 weeks
  Alpha diversity
Gut Microbiome Changes | 14 weeks
  Alpha diversity

OTHER OUTCOMES:
Safety Assessment for GI Distress | 10 weeks
  Survey based assessment
Safety Assessment for GI Distress | 14 weeks
  Survey based assessment
Facial Assessment for Redness | 10 weeks
  Via high resolution photography
Facial Assessment for Redness | 14 weeks
  Via high resolution photography

CONTACTS AND LOCATIONS:
Locations (1):
- Integrative Skin Science and Research, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No